CLINICAL TRIAL: NCT06108921
Title: Efficacy and Safety of Xylitol Nasal Irrigation After Functional Endoscopic Sinus Surgery: A Randomized Controlled Study
Brief Title: Efficacy and Safety of Xylitol Nasal Irrigation After Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CF19287A
Record Dates: First submitted 2023-10-17; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Chronic Rhinosinusitis; Postoperative Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- xylitol (Experimental): In the xylitol group, 5% xylitol solutions were first prepared by mixing two packs of 10 mg xylitol powder with 400 mL of sterile water in the container of the irrigator. Nasal irrigation was performed by using a Sanvic SH903 pulsatile irrigator (Yun-Wang Industrial Co., Tainan, Taiwan). When irrigating the nose, patients irrigated both of their nasal cavities each with 200 mL of solutions once a day. Patients performed nasal irrigations for 2 months.
  Interventions: Drug: Xylitol Powder
- saline (Placebo Comparator): In the saline group, the normal saline solution was prepared by mixing 2 packs of 1.8 mg salt powder with 400 mL of sterile water in the container of the irrigator. Nasal irrigation was performed by using a Sanvic SH903 pulsatile irrigator (Yun-Wang Industrial Co., Tainan, Taiwan). When irrigating the nose, patients irrigated both of their nasal cavities each with 200 mL of solutions once a day. Patients performed nasal irrigations for 2 months.
  Interventions: Drug: Salt Powder

INTERVENTIONS:
Drug: Xylitol Powder — The bilateral nasal cavity was irrigated by using a Sanvic SH903 pulsatile irrigator containing 400 ml of xylitol solution once a day for 2 months.
  Arms: xylitol
Drug: Salt Powder — The bilateral nasal cavity was irrigated by using a Sanvic SH903 pulsatile irrigator containing 400 ml of normal saline once a day for 2 months.
  Arms: saline

SUMMARY:
Investigators tried to evaluate the efficacy and safety of xylitol nasal irrigation as an adjuvant therapy after FESS, particularly the influence of nasal irrigation on Eustachian tube function.

DETAILED DESCRIPTION:
In this study, patients with chronic rhinosinusitis who received FESS were recruited and randomly assigned to 2 groups at one month post-surgery. Patients in the xylitol group received 400ml of 5% xylitol nasal irrigation daily for 2 months, and those in the normal saline (NS) group received 400ml of NS nasal irrigation daily for 2 months. Before FESS as well as before and after nasal irrigation, sino-nasal symptoms were assessed by a 22-item Sino-Nasal Outcome Test questionnaire and patients received endoscopic examination, nasal function tests, cytokine measurement of nasal irrigant, and bacterial culture from the middle meatus. The safety of nasal irrigation was assessed by self-reported adverse events, blood test, Eustachian Tube Dysfunction Patient Questionnaire and Eustachian tube function test. This study tried to evaluate the efficacy and safety of xylitol nasal irrigation as an adjuvant therapy after FESS, particularly the influence of nasal irrigation on Eustachian tube function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic rhinosinusitis who failed medical treatment
2. Patients underwent bilateral primary functional endoscopic sinus surgery.

Exclusion Criteria:

1. Patients with a history of immunodeficiency
2. Patients with a history of sinus surgery
3. Patients who receiving antibiotic treatment within a week before functional endoscopic sinus surgery
4. Patients with a pathological diagnosis of fungal sinusitis
5. Patients with a pathological diagnosis of sinonasal tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Taiwanese version of the 22-item Sino-Nasal Outcome Test | From before operation to 3 months after surgery
  The Taiwanese version of the 22-item Sino-Nasal Outcome Test contains 22 items of symptoms and social/emotional consequences from nasal disorder. Patients are asked to rate their problems based on how they have been over the past two weeks. Each item is graded from 0 (no problem) to 5 (as bad as it can be) according to its severity and frequency.
Self-reported adverse events | From before nasal irrigation to after 2-month nasal irrigation
  Any adverse events occurring during the 2 months period of nasal irrigation

SECONDARY OUTCOMES:
Change of the second minimal cross-sectional area of the nasal cavity | From before operation to 3 months after surgery
  The second minimal cross-sectional area of the nasal cavity was measured by acoustic rhinometry.
Change of endoscopic score | From before operation to 3 months after surgery
  The endoscopic appearances were categorized into polyps (0: no polyps; 1: polyps present within the middle meatus; 2: polyps beyond the middle meatus); nasal secretion (0: no secretion; 1: clear, thin secretion; 2: thick, purulent secretion); mucosal edema; scarring; crusting; (0: absent; 1: mild; 2: severe). The score ranged from 0 to 20 for both nostrils together.
Change of saccharine transit time | From before operation to 3 months after surgery
  The saccharine transit test involved placing saccharine granules under the head of the inferior turbinate in the more severely affected nostril. The time interval (minute) between placement of saccharine granules and sensation of sweetness in the throat was recorded.
Change of score measured by Eustachian Tube Dysfunction Patient Questionnaire | From before nasal irrigation to after 2-month nasal irrigation
  Using a 7-item Eustachian Tube Dysfunction Patient Questionnaire to evaluate Eustachian tube function
Change of Eustachian Tube function by the nine-step inflation/deflation test | From before nasal irrigation to after 2-month nasal irrigation
  Failure to alter the pressure of middle ear at least 10 daPa with swallowing during any of the steps was considered ETD (tuba1 function was 'Poor'). If the equilibration was successful (observed pressure change >10 daPa) in all steps, Eustachian tube function was considered 'Good'.

CONTACTS AND LOCATIONS:
Overall Officials: Rong-San Jiang, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, None Selected, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Outcome measures
Supporting Information: Study Protocol
Time Frame: 2 years after the end of the study
URL: https://www.vghtc.gov.tw/

REFERENCES:
- Available data/document: Study Protocol — https://www.vghtc.gov.tw/ — Study Data/Document can be requested from the PI.